CLINICAL TRIAL: NCT04302402
Title: Multi-dimensional Clinical and Pathophysiological Profiles of Patients With Functional Dyspepsia and Effect of Gut Microbiota Manipulation Using Rifaximin for Its Treatment: A Randomized Controlled Trial
Brief Title: Multi-dimensional Clinical and Pathophysiological Profiles of Patients With Functional Dyspepsia and Effect of Gut Microbiota Manipulation Using Rifaximin for Its Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Collaborators: Institute of Advanced Study in Science and Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-218-EMP-107
Record Dates: First submitted 2020-02-21; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Dyspepsia
Keywords: Pittsburgh Sleep Quality Index (PSQI); Hospital Anxiety and Depression Scale (HADS); Functional dyspepsia (FD); upper gastrointestinal (UGI)
MeSH Terms: conditions — Dyspepsia; Depression | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin (Active Comparator): Rifaximin 550mg thrice daily for 14 days Other Name: Normix
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Placebo thrice daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin has been demonstrated in multiple IBS studies, through a postulated effect on the gut microbiota, to improve the symptoms of pain and bloating, which are important symptoms in subjects with functional dyspepsia
  Other Names: Normix
  Arms: Rifaximin
Drug: Placebo — Similar looking placebo
  Arms: Placebo

SUMMARY:
Functional dyspepsia (FD) is a common condition associated with significant morbidity, healthcare expenditure, work absenteeism and productivity, and reduced quality of life. The prevalence of this condition is as high as 15% in the rural (Jaunpur district, Uttar Pradesh) and 30% of the urban (Mumbai) Indian population. Pathophysiologically, FD is an enigmatic condition that may be contributed by a variable combination of psychosocial issues like anxiety, depression, insomnia, and micro-organic issues like Helicobacter pylori infection, gastritis, duodenitis, hypersecretion of acid, degree of gastric atrophy, gastric microbiota dysbiosis. Accordingly, investigators want to study these factors among patients with FD. Rifaximin has been shown to be useful in the treatment of FD in a recent randomized controlled trial from Hong Kong. Since microbiota dysbiosis may be an important issue in FD, investigators want to treat them with rifaximin in a randomized placebo-controlled trial and repeat the parameters such as dyspepsia score, hospital Anxiety and Depression Scale (HADS) score, Pittsburgh Sleep Quality Index (PSQI). Investigators wish to study the pathogenetic mechanism of FD and evaluate baseline factors that may help to predict response to gut microbiota manipulation in these patients. Objectives: a. To study the patients with FD for gut microbiota including gastric H. pylori, gastric atrophy (by PG-1 PG-II ratio), hospital anxiety and depression score, and sleep disorders b. To see the effect of treatment of these patients with rifaximin vs. placebo in a randomized controlled trial not only for the improvement in symptoms but also for improvement in HADS score and sleep quality c. To study whether any pre-treatment factors including gut microbiota predict the response of symptoms to treatment with rifaximin.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a common clinical syndrome characterized by the presence of recurrent or chronic upper abdominal symptoms, such as epigastric pain, early satiety, and fullness, without any structural abnormalities on the upper gastrointestinal (UGI) endoscopy. FD is a heterogeneous disorder, in which different pathophysiological mechanisms underlie specific symptom patterns. It may result from a combination of visceral hypersensitivity, gastric motor dysfunction, and low-grade mucosal inflammation. Accumulating evidence including familial aggregation recently suggested that functional gastrointestinal (GI) disorders, including FD, might be contributed by genetic factors, identification of which may improve understanding of underlying pathophysiological mechanisms. Low-grade inflammation may play an important role in the pathogenesis of FD.

H. pylori infection may contribute to FD at least in a subset of patients. According to the current Rome algorithm, H. pylori infection needs to be eradicated before the diagnosis of FD is made in spite of the fact that a large proportion of patients do not improve in spite of its eradication. In addition to H. pylori, the gut microbiota is emerging to be an important player in the pathogenesis of several GI disorders including FD. In fact, several authors suggested that small bowel microbial dysbiosis, small intestinal bacterial overgrowth, and duodenal inflammation may be responsible for symptoms of FD. One of the reasons why H. pylori eradication may not give consistent results among patients with FD might be related to the fact that variable interaction between H. pylori and gut microbiota on gastric physiology might be an important player in patients with FD. Several experts suggested that variable effect H. pylori on gastric physiology may be related to its interaction with host factors and gut microbial dysbiosis might be responsible for variable efficacy of H. pylori eradication treatment in patients with FD. The role of gut microbial dysbiosis in patients with FD is supported by a recent randomized controlled trial from Hong Kong that showed rifaximin therapy targeted towards gut microbiota was useful in the treatment of patients with FD. One of the factors that may determine symptoms of FD, particularly the sub-type called epigastric pain syndrome is hypersecretion of gastric acid. Gastritis is associated both with hypochlorhydria and hyperchlorhydria; for example, antral-predominant gastritis is associated with hyperchlorhydria and body-predominant gastritis is associated with hypochlorhydria. Pepsinogen I and II ratio is a non-invasive method to assess the topography of gastritis, such as antral or body predominant. Pepsinogen is the inactive precursor of the gastric proteolytic enzyme pepsin. Human pepsinogen comprises two isoenzymes, pepsinogen I (or A) and pepsinogen II (or C). Pepsinogen I (PG-I) is secreted mainly by chief cells of fundic mucosa, whereas pepsinogen II (PG-II) is also secreted by pyloric glands and proximal duodenal mucosa. While serum levels of PG-I correlate with levels of acid secretion, PG-II shows an inverse relationship. Therefore, the PG-I/PG-II ratio is a useful tool to evaluate gastric acid secretion, gastritis, and intestinal metaplasia. Gastrin secretion is regulated by a negative feedback mechanism looped with acid secretion. In fact, the patients with functional gastrointestinal disorders (FGIDs) were earlier thought to be psychogenic in origin; this understanding might have resulted in the development of a belief among treating physicians/gastroenterologists that these patients are rather neurotic, apprehensive individual feigning an illness. Such erroneous belief might have resulted in disservice to these patients. However, recently accumulating evidence suggests that patients with FGIDs have several pathophysiological abnormalities in the gastrointestinal (GI) tract that might not be visualized by conventional investigations such as upper GI endoscopy but are often visible with more sophisticated tests including molecular techniques. Hence, we proposed that these disorders be called micro-organic disorders. In fact, experts in Rome Foundation in the Rome IV algorithm suggested that these disorders need to be considered as disorders of "gut-brain interaction" rather than "brain-gut interaction" reinforcing the importance of the peripheral rather than central mechanisms in the pathogenesis. Rome IV also suggests that in clinical practice, a multi-dimensional clinical profile of the FGIDs (which include the categorical diagnosis, subtype, severity, psychological factors, and physiological factors including biomarkers) needs to be uncovered before further treatment of these patients. This is a paradigm shift in understanding pathogenesis and treatment of the FGIDs including FD but needs more evidence particularly from tropical and sub-tropical areas of the World. Hence, the clinical and scientific importance of the proposed study can't be over-estimated. Functional dyspepsia (FD) is an enigmatic condition that may be contributed by a variable combination of psychosocial issues like anxiety, depression, insomnia, and micro-organic issues like Helicobacter pylori infection, gastritis, duodenitis, hypersecretion of acid, degree of gastric atrophy, gastric microbiota dysbiosis. Accordingly, we aimed to study these factors among patients with FD. Rifaximin has been shown to be useful in the treatment of FD in a recent randomized control trial from Hong Kong. Since microbiota dysbiosis may be an important issue in FD, we planned to treat them with rifaximin in a randomized placebo-controlled trial and repeat the parameters such as dyspepsia score, hospital Anxiety and Depression Scale (HADS) score, Pittsburgh Sleep Quality Index (PSQI). We wish to study the pathogenetic mechanism of FD and evaluate baseline factors that may help to predict response to gut microbiota manipulation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* FD diagnosis by ROME IV criteria (one or more of bothersome symptoms like postprandial fullness, early satiation, epigastric pain, and epigastric burning. It must include criteria for postprandial distress syndrome and epigastric pain syndrome for the last 3 months with symptom onset at least 6 months before diagnosis and no evidence of structural disease, including upper endoscopy).
* No organic disease on upper gastrointestinal endoscopy and ultrasound.
* Currently, not on any active therapy during the last two months.
* No previous history of Helicobacter pylori eradication.
* No antibiotic therapy within the last month.
* Not received proton pump inhibitors for a minimum of 4 weeks prior to study enrollment.

Exclusion Criteria:

* Presence of alarm symptoms such as GI bleeding, unexplained iron deficiency anemia, unintentional weight loss, palpable abdominal mass, family history of colon or stomach cancer or symptom onset ≥50 years of age and not yet screened for colon cancer, or sudden/acute onset of a new change in bowel habit)
* No proper informed consent.
* Endoscopic treatment for gastroesophageal reflux.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in composition of gut microbiota | Baseline upto 6 months
  To study changes from baseline in composition of gut microbiota including gastric H. pylori, gastric atrophy (PG-I, PG-II ratio
Hospital anxiety and depression score | Baseline upto 6 months
  Number of items in the questionnaire reflects anxiety and depression. Each item had been answered by the patient on a four point (0-3) response category and the possible scores ranged from 0-21 for depression (0-7 score indicates normal range, 8-10 indicates 'borderline abnormal or borderline case' and a score of 11 or higher indicates 'abnormal case'.

SECONDARY OUTCOMES:
Sleep quality index score | Baseline upto 6 months
  Self-reported usual sleep habits for the majority of days and nights during the past month only. The 19 self-rated and 5 non-self rated questions combined to form seven component scores, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Uday C Ghoshal, Principal Investigator — Medical council of India, Association of Indian Universities
Locations (2):
- India (2):
  - Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No
This study will be conducted in the Department of Gastroenterology, in inter-institutional collaboration with Dr. Mojibur R. Khan (Gut Microbiome expert) from Life Science Division, Institute of Advanced Study in Science and Technology (IASST) and in inter-departmental collaborations with the department of Microbiology having patients with clinical suspicion with FD and facility for laboratory works.

REFERENCES:
- [Result] Li X, Cao Y, Wong RK, Ho KY, Wilder-Smith CH. Visceral and somatic sensory function in functional dyspepsia. Neurogastroenterol Motil. 2013 Mar;25(3):246-53, e165. doi: 10.1111/nmo.12044. Epub 2012 Nov 21. PMID 23171089
- [Result] Sebastian-Domingo JJ. [Integrative medicine in the management of functional dyspepsia. Role of the herbal preparation STW5]. Gastroenterol Hepatol. 2014 Apr;37(4):256-61. doi: 10.1016/j.gastrohep.2013.10.001. Epub 2013 Dec 5. Spanish. PMID 24314790